CLINICAL TRIAL: NCT00170846
Title: Assessment of Everolimus in Addition to Calcineurin Inhibitors Reduction in Maintenance Renal Transplant Recipients
Brief Title: ASCERTAIN: Assessment of Everolimus in Addition to Calcineurin Inhibitor Reduction in the Maintenance of Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2413
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2011-03

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, everolimus, calcineurin inhibitors, GFR
MeSH Terms: interventions — Everolimus; Calcineurin Inhibitors; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A: No RAD (Active Comparator): Calcineurin Inhibitors (CNI) ± Mycophenolate Acid (MPA)/Azathioprine (AZA) ± Steroids
  Interventions: Drug: Calcineurin Inhibitors (CNI); Drug: Mycophenolate acid (MPA)/Azathioprine (AZA); Drug: Steroids
- Group B : CNI Withdrawal (Experimental): Initiation of everolimus (8-12 ng/mL) with discontinuation of CNI. Everolimus(RAD001) 4 mg initial daily dose.
  Interventions: Drug: Everolimus (RAD001); Drug: Mycophenolate acid (MPA)/Azathioprine (AZA); Drug: Steroids
- Group C: CNI Reduction (Experimental): Initiation of everolimus (3-8 ng/mL) with reduction by 70-90% in CNI blood levels. Everolimus (RAD001) 3 mg initial daily dose.
  Interventions: Drug: Everolimus (RAD001); Drug: Calcineurin Inhibitors (CNI); Drug: Mycophenolate acid (MPA)/Azathioprine (AZA); Drug: Steroids

INTERVENTIONS:
Drug: Everolimus (RAD001)
  Arms: Group B : CNI Withdrawal; Group C: CNI Reduction
Drug: Calcineurin Inhibitors (CNI)
  Arms: Group A: No RAD; Group C: CNI Reduction
Drug: Mycophenolate acid (MPA)/Azathioprine (AZA)
Drug: Steroids

SUMMARY:
The study is designed to evaluate whether the initiation of everolimus together with the reduction or discontinuation of calcineurin inhibitors (CNIs) will improve graft function in the maintenance of renal transplant recipients with renal impairment by reducing the progression of chronic allograft nephropathy. The development of atherosclerosis in the native arteries of the patients will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient at least 18 years of age.
* Patient who has undergone a primary or secondary renal transplant 12-96 months ago from a living related or unrelated donor or a cadaveric donor.
* Patient receiving cyclosporine microemulsion with a C2-h level ≥ 400 ng/mL or tacrolimus with a C0-h level ≥ 4 ng/mL with or without mycophenolic acid or azathioprine plus or minus steroids.
* The immunosuppressive regimen must remain unchanged within the last 3 months.
* Patient with renal impairment defined as GFR between 30 and 70 mL/min/1.73 m^2 by Cockcroft-Gault formula.

Exclusion Criteria:

* Patient who is recipient of multiple organ transplants.
* Patient with protein/creatinine ratio ≥ 150 (mg/mmol).
* Patient with a treated acute rejection episode within the last 3 months.
* Patient with any past or present BK-polyomavirus nephropathy.
* Patient with de novo or recurrent glomerular nephritis.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2005-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B : CNI Withdrawal: Initiation of everolimus (8-12 ng/mL) with discontinuation of CNI. Everolimus (RAD001) 4 mg initial daily dose.
Period: Overall Study
Arm/Group | Group A: No RAD | Group B : CNI Withdrawal | Group C: CNI Reduction
Started | 123 | 127 | 144
Completed | 112 | 108 | 131
Not Completed | 11 | 19 | 13
Not completed — Subject withdrew Informed Consent | 5 | 12 | 8
Not completed — Lost to Follow-up | 6 | 3 | 2
Not completed — Death | 0 | 3 | 3
Not completed — Reason Missing | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: No RAD | Group B : CNI Withdrawal | Group C: CNI Reduction | Total
Number analyzed (Participants) | 123 | 127 | 144 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (12.18) | 49.4 (11.81) | 49.7 (12.95) | 49.1 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 53 | 135
  Male | 82 | 86 | 91 | 259
Time since transplantation [Mean (Standard Deviation); unit: years] | 5.8 (4.14) | 5.4 (4.28) | 5.4 (3.99) | 5.6 (4.13)

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Assessed by Measured GFR (mGFR)
Description: The acceptable methods for GFR measurement were Chromium 51-Ethylenediaminetetra acetic acid (Cr-EDTA), Technetium 99-Diethylenetriaminepentacetic acid (Tc-DTPA), Iohexol clearance Inuline clearance and Iothalamate clearance. The method should have been consistent for a given patient at every time point.
Time Frame: 24 months
Population: The modified ITT population included all ITT patients who had mGFR or calculated GFR (cGFR) at Month 24 based on all values including those collected after discontinuation of study medication.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Group A: No RAD | Group B : CNI Withdrawal | Group C: CNI Reduction
Number analyzed (Participants) | 103 | 94 | 109
mL/min/1.73m^2 | 46.02 (20.358) | 48.00 (22.033) | 46.60 (21.079)
Statistical Analysis 1: Comparison: Group A: No RAD vs Group B : CNI Withdrawal; Test type: Superiority or Other; p = 0.6332, ANCOVA; Difference in LS means = 1.1241, 95% CI 2-sided [-3.5077 to 5.7559]
Statistical Analysis 2: Comparison: Group A: No RAD vs Group C: CNI Reduction; Test type: Superiority or Other; p = 0.7943, ANCOVA; Difference in LS means = 0.5933, 95% CI 2-sided [-3.8815 to 5.0682]

2. Post Hoc Outcome: Change in mGFR by Baseline Calculated Creatinine Clearance (Cockcroft-Gault Formula)
Description: Cockcroft-Gault formula (CrCl):
  Creatinine Clearance [mL/min] = CrCl (males) = (140 - A) * W / (72 * C) (males), CrCl (females) = CrCl (males) * 0.85,
  Where:
  * A is age [years]
  * W is body weight [kg]
  * C is the serum concentration of creatinine [mg/dL]
Time Frame: Baseline and 24 months
Population: Per Protocol Population. The per-protocol (PP) population consisted of the ITT patients excluding those patients with major protocol deviations and those patients who were not able to initiate their randomized regimens as scheduled.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group A: No RAD | Group B : CNI Withdrawal | Group C: CNI Reduction
Number analyzed (Participants) | 112 | 110 | 124
mL/min
  Baseline CrCl(CG) ≤ 50 :(n= 32, 28, 32):- Change | 1.55 (12.833) | -5.75 (14.712) | 0.82 (19.445)
  Baseline CrCl(CG) > 50 : (n=31, 29, 39):-Change | -2.55 (19.562) | 7.32 (21.051) | -0.24 (17.551)

3. Secondary Outcome: Number of Participants With Safety Parameters
Description: The selected safety parameters (such as hypertension, hyperlipidemia, diabetes mellitus, anemia, malignancies ) were derived based on adverse events preferred terms defined in the analysis plan.
Time Frame: 24 months
Population: Safety Population. The Safety Population consisted of all randomized patients who received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Group A: No RAD | Group B : CNI Withdrawal | Group C: CNI Reduction
Number analyzed (Participants) | 123 | 127 | 144
Participants
  Hypertension, Yes | 6 | 13 | 9
  Hypertension, No | 117 | 114 | 135
  Hyperlipidemia, Yes | 6 | 18 | 11
  Hyperlipidemia, No | 117 | 109 | 133
  Diabetes mellitus, Yes | 4 | 6 | 7
  Diabetes mellitus, No | 119 | 121 | 137
  Anemia, Yes | 25 | 45 | 46
  Anemia, No | 98 | 82 | 98
  Malignancies, Yes | 7 | 9 | 11
  Malignancies, No | 116 | 118 | 133

ADVERSE EVENTS:
Arm/Group | Group A: No RAD | Group B : CNI Withdrawal | Group C: CNI Reduction
Serious Adverse Events (participants affected / at risk) | 52/123 | 72/127 | 78/144
Other Adverse Events (participants affected / at risk) | 97/123 | 116/127 | 126/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: No RAD (N=123) | Group B : CNI Withdrawal (N=127) | Group C: CNI Reduction (N=144)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 3
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 12
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5 | 4
Asthenia (General disorders) | 0 | 0 | 3
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 3
Pyrexia (General disorders) | 1 | 4 | 11
Sudden death (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 2
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Abscess fungal (Infections and infestations) | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Carbuncle (Infections and infestations) | 0 | 0 | 1
Cardiac infection (Infections and infestations) | 0 | 0 | 1
Catheter sepsis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 3 | 4
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Endocarditis (Infections and infestations) | 0 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 4 | 6
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 1
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 2
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Mucormycosis (Infections and infestations) | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oophoritis (Infections and infestations) | 0 | 0 | 2
Oral infection (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 5
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Salmonella sepsis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 3 | 2
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 2
Tuberculosis bladder (Infections and infestations) | 1 | 0 | 0
Tuberculosis of genitourinary system (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 1
Urethral abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 5 | 10
Urosepsis (Infections and infestations) | 0 | 1 | 1
Varicella (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 2 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 3 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 2 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal graft loss (Injury, poisoning and procedural complications) | 4 | 3 | 9
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 7 | 7 | 4
Blood folate decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 0
Blood uric acid increased (Investigations) | 2 | 0 | 0
Protein urine (Investigations) | 0 | 0 | 1
Tuberculin test positive (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1
Vitamin B12 decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myositis ossificans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 4
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrectasia (Renal and urinary disorders) | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 3 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 3 | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: No RAD (N=123) | Group B : CNI Withdrawal (N=127) | Group C: CNI Reduction (N=144)
Anaemia (Blood and lymphatic system disorders) | 22 | 42 | 40
Leukopenia (Blood and lymphatic system disorders) | 5 | 10 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 10 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 22 | 9
Diarrhoea (Gastrointestinal disorders) | 20 | 36 | 30
Mouth ulceration (Gastrointestinal disorders) | 1 | 15 | 8
Nausea (Gastrointestinal disorders) | 7 | 9 | 7
Vomiting (Gastrointestinal disorders) | 7 | 7 | 9
Oedema (General disorders) | 0 | 8 | 6
Oedema peripheral (General disorders) | 12 | 33 | 37
Pyrexia (General disorders) | 6 | 15 | 16
Bronchitis (Infections and infestations) | 7 | 6 | 6
Nasopharyngitis (Infections and infestations) | 8 | 9 | 13
Upper respiratory tract infection (Infections and infestations) | 16 | 11 | 15
Urinary tract infection (Infections and infestations) | 10 | 20 | 18
Blood creatine phosphokinase increased (Investigations) | 2 | 7 | 3
Blood creatinine increased (Investigations) | 15 | 11 | 10
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 3
Gout (Metabolism and nutrition disorders) | 7 | 4 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 18 | 24
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 18 | 11
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 6 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 12 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 3 | 11
Dizziness (Nervous system disorders) | 5 | 4 | 9
Headache (Nervous system disorders) | 5 | 7 | 12
Proteinuria (Renal and urinary disorders) | 11 | 18 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 18 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9
Acne (Skin and subcutaneous tissue disorders) | 1 | 16 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 20 | 12
Hypertension (Vascular disorders) | 5 | 12 | 8
Hypotension (Vascular disorders) | 1 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.